CLINICAL TRIAL: NCT06447896
Title: A Open-label, Randomised, Paired Design, Multicenter Study of a Cardiovascular Autonomic Nervous Function Multi-Parameter Evaluation System With Intelligent Human-Machine Interaction for Assessing Cardiovascular Autonomic Neuropathy
Brief Title: Clinical Validation of a Cardiovascular Autonomic Nervous Function Multi-Parameter Evaluation System
Acronym: CARTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: REEM (Shenzhen) Healthcare Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CARTS20210908
Record Dates: First submitted 2024-05-28; First posted 2024-06-07 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Cardiovascular Autonomic Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): In the experimental arm, the Cardiovascular Autonomic Nervous Function Multi-Parameter Evaluation System (Model: R6000, REEM (Shenzhen) Healthcare Co., Ltd) is used for both cardiovascular autonomic reflex tests (CARTs) and heart rate variability (HRV) analysis.
  Interventions: Device: Cardiovascular Autonomic Nervous Function Multi-Parameter Evaluation System (Model: R6000)
- Arm B (Active Comparator): In the active comparator arm, conventional method of CARTs and HRV analysis using a commercially available ambulatory holter station are conducted as control.
  Interventions: Diagnostic Test: Conventional method of CARTs; Device: Ambulatory holter station Model i12 plus

INTERVENTIONS:
Device: Cardiovascular Autonomic Nervous Function Multi-Parameter Evaluation System (Model: R6000) — Cardiovascular autonomic reflex tests (CARTs) and heart rate variability analysis (HRV) are conducted with Cardiovascular Autonomic Nervous Function Multi-Parameter Evaluation System (Model: R6000). CARTs include five standardized tests, which are heart rate response to lying-to-standing, Valsalva maneuver, deep breathing, and blood pressure response to lying-to-standing and sustained isometric handgrip. These series of movements act as "standardized stimuli" to trigger hemodynamic changes in the body, altering vagal and sympathetic activity through mechanisms such as the baroreflex, thereby producing changes in heart rate and blood pressure. The sensor-monitoring interactive design of the device ensures the standardization of these maneuvers.
  Arms: Arm A
Diagnostic Test: Conventional method of CARTs — Conventional method are conduced using blood pressure kit with manual sphygmomanometer and ECG machine. Conventional method and the investigated device are used simultaneously to record electrocardiograms. Conventional blood pressure taking are carried out in sequence with the investigated device. CARTs results from the conventional method are used as control.
  Arms: Arm B
Device: Ambulatory holter station Model i12 plus — Model i12 plus (manufactured by RENCARE) is an ambulatory holter station, which was approved by the Center for Medical Device Evaluation (CMDE), China National Medical Products Association (NMPA). It can analyze electrocardiogram and generate HRV indices, which include SDNN, RMSSD, NN50, pNN50, triangular index, average RR, deceleration capacity (DC), deceleration runs (DRs), VLF, LF, HF, LF/HF, and total power. Model i12 plus is used to analyzed the same ECG signals as the investigated device.
  Arms: Arm B

SUMMARY:
This is a open-label, randomized, paired design, multicenter study of the Cardiovascular Autonomic Nervous Function Multi-Parameter Evaluation System (R6000) for evaluating cardiovascular autonomic neuropathy. R6000 is novel intellectual diagnostic device for cardiovascular autonomic reflex tests and heart rate variability analysis. A total of 85 subjects will be enrolled in trial Ⅰ and 150 subjects will be enrolled in trial Ⅱ. In trial Ⅰ, subjects will be randomized to two groups, one of which will receive test by the tested device first and the other one will be tested by conventional blood pressure kit. The primary objective of this clinical trial is to evaluate the effectiveness of the Cardiovascular Autonomic Nervous Function Multi-Parameter Evaluation System. The secondary objective is to evaluate the safety of the cardiovascular autonomic testing system and stability.

DETAILED DESCRIPTION:
Trial I Tested device: Cardiovascular Autonomic Nervous Function Multi-Parameter Evaluation System (R6000). Control: Conventional blood pressure kit. Goal: To assess the consistency between the tested device and the conventional method in measuring blood pressure.

Trial IIa Tested device: Cardiovascular Autonomic Nervous Function Multi-Parameter Evaluation System (R6000). Control: Ambulatory holter station. Goal: To assess the consistency between the tested device and the conventional devices in measuring heart rate variability (HRV).

Trial IIb Tested device: Cardiovascular Autonomic Nervous Function Multi-Parameter Evaluation System (R6000). Control: Manual method with digital ECG machine, stethoscope and sphygmomanometer. Goal: To assess the consistency between the tested device and the manual method in determining cardiovascular autonomic neuropathy (CAN).

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 or over, regardless of gender
* Voluntary membership to participate in the study and signing the Informed Consent Form.

Exclusion Criteria:

* For part I:

  • Unable to cooperate with the examination.
* For part II:

  * Ophthalmic examination within the past 1 month showed proliferative retinopathy, retinal detachment, fundus hemorrhage or presence of known history of illness described above;
  * Known history of glaucoma or ophthalmic examination within the past 1 month suggests glaucoma;
  * Poor control of hypertension (sedentary systolic blood pressure ≥ 160mmHg or diastolic blood pressure ≥100mmHg);
  * Known history of arrhythmia (except occasional premature beats), history of acute coronary syndrome within three months before signing the informed consent form;
  * In a state of stress such as infection and surgery; Be in the acute or unstable phase of any disease;
  * Pregnant women;
  * Unable to cooperate with the examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2011-03-11 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
The diagnostic accuracy of the tested device versus manual method for the diagnosis of cardiovascular autonomic neuropathy (CAN). | up to 6 months
  Cohen's kappa coefficient will be used to assess the consistency between the tested device and the manual method in determining CAN status (positive or negative). The assessment will be conducted in part IIb.

SECONDARY OUTCOMES:
The accuracy of the tested device versus conventional blood pressure kit with Korotkoff auscultatory technique for measuring blood pressure. | up to 6 months
  In part I, secondary outcome measures include the average difference and standard deviation of systolic and diastolic blood pressure values obtained using the tested device and the conventional blood pressure kit with Korotkoff auscultatory technique.
The accuracy of the tested device versus the control device for measuring HRV. | up to 6 months
  In part IIa, secondary outcome measures involve a comparative analysis of HRV indices obtained using the tested device and the control device.

IPD SHARING:
Plan to Share IPD: No